CLINICAL TRIAL: NCT00673751
Title: GLP-2 Mediated Increased SMA Blood Flow in Patients With Short Bowel Syndrome
Brief Title: Effect of the Enteric Hormone Glucagon-Like Peptide (GLP-2) on the Intestinal Blood Flow in Patients With Short Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Lasse Bremholm, Dept. of gastroenterology, Glostrup Hospital, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: H-A-2008-032
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Short Bowel Syndrome
Keywords: mesenteric blood flow; GLP-2; short bowel syndrome; Glucagon-Like Peptide 2
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): subcutaneous isotonic saline
  Interventions: Drug: Placebo
- 1 (Active Comparator): subcutaneous GLP-2
  Interventions: Drug: GLP-2

INTERVENTIONS:
Drug: GLP-2 — 450 nmol subcutaneous
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The aim of the study is to investigate the effect of the enteric hormone Glucagon-like Peptide (GLP-2) on patients with short bowel syndrome

DETAILED DESCRIPTION:
previous studies have shown that GLP-2 increases mesenteric blow flow, we wish to examine the effect of subcutaneus GLP-2 on patients with short bowl syndrome. The patients will single blinded been given 450 nmol GLP-2 and isotonic saline in order to act as their own reference.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnose of short bowel syndrome 4 month of stable fase

Exclusion Criteria:

* activity in IBD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Glostrup University Hospital, Glostrup Municipality, Capital Region, Denmark